CLINICAL TRIAL: NCT03931057
Title: The Use of ADV6209 for Premedication in Pediatric Anesthesia: a Controlled, Randomized, Double Blinded Study
Brief Title: The Use of ADV6209 for Premedication in Pediatric Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Peter Marhofer, Clinical Professor, MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1.4-22.07.2019
Record Dates: First submitted 2019-04-23; First posted 2019-04-29 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Preanesthetic Medication
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Intervention Model Description: A controlled, randomized, double blinded study Study group 1 (40 children) ADV6209 0.25 mg/kg p.o. Study group 2 (40 children) Midazolam (in orange flavoured syrup) 0.25 mg/kg p.o.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADV6209 (Experimental): ADV6209 (= gamma-cyclodextrin-Midazolam) 0.25 mg/kg p.o. once 30 min. before anesthesia
  Interventions: Drug: ADV6209 (=gamma-cyclodextrin-Midazolam)
- Midazolam (Active Comparator): Midazolam (in orange flavored syrup) 0.25 mg/kg p.o. once 30 min. before anesthesia
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: ADV6209 (=gamma-cyclodextrin-Midazolam) — 30 min. before anesthesia children have to swallow the anxiolytic drug (ADV6209)
  Other Names: Ozalin (registered Tradename)
  Arms: ADV6209
Drug: Midazolam — 30 min. before anesthesia children have to swallow the anxiolytic drug Midazolam
  Other Names: Dormicum (Tradename)
  Arms: Midazolam

SUMMARY:
To evaluate the effect of ADV6209, a new oral Midazolam formulation, on preoperative anxiety and sedation levels in paediatric anaesthesia Primary Objective: Sedation score (mYPAS) 30 min after administration of the premedication drug Secondary Objective: Acceptance of anaesthesia mask induction Acceptance of oral administration of the premedication drug

DETAILED DESCRIPTION:
Premedication represents an important part in the perioperative management of children and is used to reduce pre-operative stress as well as to facilitate induction of inhaled anaesthesia. Midazolam is the drug most often used for premedication in infants and children because it provides good sedation, anxiolytic and amnestic effects and few side effects. Oral intake of the drug is the most preferred route of administration by paediatric patients, whereas the majority of existing oral Midazolam solutions involve the use of i.v. Midazolam formulation given orally, unregistered or off-label. Moreover i.v. Midazolam solutions are often not well accepted by children because of their bitter taste. Considering the lack of available oral medications for moderate sedation in children in most European countries, ADV6209, an innovative 0.2% (w/v) oral solution of Midazolam for children from six months of age, was developed. The formation of a γ-Cyclodextrin -Midazolam complex, representing a new chemical formula, was used to improve the solubility and the palatability of the Midazolam formulation. A pharmacokinetic (PK) study has been executed in adults, children and adolescents, whereas ADV6209 showed improvements to current extemporaneous oral solutions of midazolam (EOM) preparations in terms of taste and easiness of use while presenting a similar PK profile. Satisfying sedation, measured with the Observer Assessment of Alertness/Sedation Scale (OAA score / S≤17) was observed in 78.4% of paediatric patients 30 minutes after ADV6209 administration. Anxiety score (modified Yale Preoperative Anxiety Scale - mYPAS) was decreased by 18.3% on average over baseline, 30 minutes after ADV6209 with a more pronounced effect in the youngest children who were also the most anxious prior to administration of the drug. In general the treatment was well accepted by all children and did not induce more crying and nausea / vomiting than before Midazolam. ADV6209 seems a very promising premedication drug. It has been licensed by the EU regulatory authorities to become the first licensed paediatric sedative in the EU (September 2018). It may help to avoid unregistered and off label use of EOM. Consequently, we want to evaluate the efficacy and safety of ADV6209 on preoperative anxiety and sedation levels in paediatric anaesthesia in daily clinical routine in this randomized, controlled, double blinded study.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 and 2 children from 2-8 years scheduled for elective surgical or diagnostic procedures, where premedication would be used in clinical routine
* Signed written parental informed consent prior to inclusion in the study

Exclusion Criteria:

* ASA 3-5
* Allergy against the study drug
* Participation in another clinical study investigating another IMP within one month prior to screening
* Other objections to study participation in the opinion of the investigator
* Parent's or legal guardian's refusal of participation of the child

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2021-09-17 (Actual)

PRIMARY OUTCOMES:
Change from baseline of the sedation score (modified Yale Preoperative Anxiety Scale - mYPAS-short form) at 30 minutes after administration of the premedication drug | The level of sedation 1 minute before the premedication will be graded and compared to the level of sedation 30 minutes after the oral administration of the drug
  The mYPAS-SF consists of four items (activity, vocalizations, emotional expressivity and state of apparent arousal). Each domain consists of Likert-type response options reflecting behaviours. Children's behaviour is rated from 1 to 4 or 1 to 6 (depending on the domain), with higher numbers indicating the highest severity within that domain

SECONDARY OUTCOMES:
Acceptance of oral administration of the premedication drugs | Will be evaluated, when the children swallow the premedication drug - 30 minutes before the induction of anaesthesia
  Observers record the child's acceptance of the orange-flavoured γ-Cyclodextrin -Midazolam (Ozalin®) (intervention group) or the Midazolam in orange - flavoured syrup (control group) according to the following graduation immediately after administration of the study drug: (1) The child accepts readily, (2) the child accepts with facial grimace, (3) the child accepts with verbal complaint or (4) the child rejects entirely or spits out almost/or all of the dose.
Acceptance of anaesthesia mask induction | Will be evaluated, when anaesthesia is induced with the anesthesia mask - 30 minutes after the premedication
  Mask Acceptance Score: A four-point mask-induction score will be used to determine the quality of induction of narcosis via face mask as follows: (1) Very good, immediate acceptance of the face mask, (2) good, slight resistance, (3) moderate, struggle against face mask and (4) difficult, moderate force necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Marhofer, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Dept. of Anesthesia, Intensive Care Medicine and Pain Medicine, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kain ZN, Mayes LC, Cicchetti DV, Bagnall AL, Finley JD, Hofstadter MB. The Yale Preoperative Anxiety Scale: how does it compare with a "gold standard"? Anesth Analg. 1997 Oct;85(4):783-8. doi: 10.1097/00000539-199710000-00012. PMID 9322455
- [Background] Kain ZN, Caldwell-Andrews AA, Krivutza DM, Weinberg ME, Wang SM, Gaal D. Trends in the practice of parental presence during induction of anesthesia and the use of preoperative sedative premedication in the United States, 1995-2002: results of a follow-up national survey. Anesth Analg. 2004 May;98(5):1252-9, table of contents. doi: 10.1213/01.ane.0000111183.38618.d8. PMID 15105196
- [Background] Marcon F, Mathiron D, Pilard S, Lemaire-Hurtel AS, Dubaele JM, Djedaini-Pilard F. Development and formulation of a 0.2% oral solution of midazolam containing gamma-cyclodextrin. Int J Pharm. 2009 Sep 11;379(2):244-50. doi: 10.1016/j.ijpharm.2009.05.029. Epub 2009 May 23. PMID 19467307
- [Background] Cuzzocrea F, Gugliandolo MC, Larcan R, Romeo C, Turiaco N, Dominici T. A psychological preoperative program: effects on anxiety and cooperative behaviors. Paediatr Anaesth. 2013 Feb;23(2):139-43. doi: 10.1111/pan.12100. PMID 23289773
- [Background] Davidson AJ, Shrivastava PP, Jamsen K, Huang GH, Czarnecki C, Gibson MA, Stewart SA, Stargatt R. Risk factors for anxiety at induction of anesthesia in children: a prospective cohort study. Paediatr Anaesth. 2006 Sep;16(9):919-27. doi: 10.1111/j.1460-9592.2006.01904.x. PMID 16918652
- [Background] Fortier MA, MacLaren JE, Martin SR, Perret-Karimi D, Kain ZN. Pediatric pain after ambulatory surgery: where's the medication? Pediatrics. 2009 Oct;124(4):e588-95. doi: 10.1542/peds.2008-3529. Epub 2009 Sep 7. PMID 19736260
- [Background] Fortier MA, Del Rosario AM, Martin SR, Kain ZN. Perioperative anxiety in children. Paediatr Anaesth. 2010 Apr;20(4):318-22. doi: 10.1111/j.1460-9592.2010.03263.x. Epub 2010 Feb 23. PMID 20199609
- [Background] Marcon F, Guittet C, Manso MA, Burton I, Granier LA, Jacqmin P, Dupont H. Population pharmacokinetic evaluation of ADV6209, an innovative oral solution of midazolam containing cyclodextrin. Eur J Pharm Sci. 2018 Mar 1;114:46-54. doi: 10.1016/j.ejps.2017.11.030. Epub 2017 Dec 5. PMID 29203151
- [Background] Huet A, Lucas-Polomeni MM, Robert JC, Sixou JL, Wodey E. Hypnosis and dental anesthesia in children: a prospective controlled study. Int J Clin Exp Hypn. 2011 Oct-Dec;59(4):424-40. doi: 10.1080/00207144.2011.594740. PMID 21867378
- [Background] Weldon BC, Bell M, Craddock T. The effect of caudal analgesia on emergence agitation in children after sevoflurane versus halothane anesthesia. Anesth Analg. 2004 Feb;98(2):321-326. doi: 10.1213/01.ANE.0000096004.96603.08. PMID 14742362
- [Background] Schulz KF, Altman DG, Moher D, Fergusson D. CONSORT 2010 changes and testing blindness in RCTs. Lancet. 2010 Apr 3;375(9721):1144-6. doi: 10.1016/S0140-6736(10)60413-8. Epub 2010 Mar 24. No abstract available. PMID 20338625